CLINICAL TRIAL: NCT06647602
Title: Thyroid Hormone Replacement After Radio Iodine: Value and Efficacy
Acronym: THRIVE
Status: Not yet recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 11432; 2024-511668-10-00 (EU CTIS Number)
Record Dates: First submitted 2024-06-11; First posted 2024-10-18 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Differentiated Thyroid Cancer; Thyroid Cancer; Levothyroxine; Liothyronine; Thyroid Hormones
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Thyroxine; Triiodothyronine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples from venapuncture
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- TH-combination cohort: L-T4+L-T3 combination according to local protocol.
  Interventions: Drug: Cytomel (liothyronine)
- Levothyroxine cohort: L-T4 monotherapy according to local protocol.
  Interventions: Drug: Euthyrox (levothyroxine)

INTERVENTIONS:
Drug: Euthyrox (levothyroxine) — Euthyrox (levothyroxine sodium tablets; L-T4) is a thyromimetic synthetic drug identical to T4. Patients will recieve levothyroxine (euthyrox) in a dose of 2 μg × kg body weight / day.
  Groups: Levothyroxine cohort
Drug: Cytomel (liothyronine) — Cytomel (liothyronine sodium tablets; L-T3) is a thyromimetic synthetic drug identical to T3.
  The patients in this cohort recieve L-T4+L-T3 combination therapy. The L-T4 dose will be 2 μg × kg body weight / day, equal to the dose in the other interventional arm. L-T3 will be added twice daily from the first day of combination treatment, in dosages gradually decreasing from 25 ug 2/day to 5 ug 2/day over a time span of 3 weeks after which L-T3 is stopped.
  Groups: TH-combination cohort

SUMMARY:
This study will be a multicentre prospective cohort study on TH-substitution after thyroid hormone withdrawal preceding radioiodine treatment.

DETAILED DESCRIPTION:
While treatment with L-T4 after TH-withdrawal is widely used in DTC patients to suppress TSH and improve hypothyroid symptoms, the value of L-T3 addition in initiation of TH treatment has not been evaluated in this context. Lifelong monotherapy with L-T3 should not be preferred over L-T4 yet, short-term use of L-T3 to initiate TH-supplementation can be safely implemented. We hypothesize that initial treatment with L-T4+L-T3 combination treatment can have a more direct effect on TSH-levels and earlier relieve of hypothyroid symptoms resulting in a better QoL. We will conduct a prospective cohort study comparing the initiation of TH-supplementation after TH-withdrawal in two cohorts of DTC patients: patients receiving L-T4+LT3 with a gradually decrease of L-T3 dose in time, and patients receiving L-T4 only. We will compare potency to suppress TSH, effect on QoL and effects on thyroid- and cardiovascular parameters. Patients (18-75 years) diagnosed with high-risk DTC after TH-withdrawal will be eligible for inclusion. The primary objective is to compare the proportion of patients reaching target TSH-levels after two weeks of substitution with L-T3 or L-T4.

Secondary objectives are to compare the effects of L-T4+L-T3 or L-T4 in the first 3 months of treatment on serum thyroid parameters TSH and Tg, quality of life, and cardiovascular parameters

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed DTC (papillary thyroid carcinoma, follicular thyroid carcinoma, oncocytic thyroid carcinoma)
* Classified as high-risk DTC according to the ATA guidelines or, patients for whom the risk of a recurrence is estimated to be higher based on clinical features (assessed by their treating physician).
* Prepared for RAI-therapy with TH-withdrawal
* Patients must be fit to adhere to the study protocol
* Patients must be able to read and understand the Dutch language

Exclusion Criteria:

* Pregnancy
* Patients with comorbidities, such as severe heart failure, (poorly controlled) atrial fibrillation, of which the treating physician decides that L-T3 is unsuitable.
* Conditions or drugs interfering with thyroid hormone uptake:
* Patients with a history of atrophic gastritis
* Patients using proton-pomp inhibitors

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include patients with a histologically confirmed high-risk DTC, men and women aged 18-75 years. Patients have to be prepared to RAI with TH-withdrawal and treated according to the ATA guidelines.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
TSH after two weeks of TH substitution | Before and after 2 weeks of TH-substitution
  The percentage of patients reaching target TSH (<0.5 mU/L) after two weeks of L-T3+L-T4 substitution compared to patients with L-T4-substitution.

SECONDARY OUTCOMES:
TSH (mU/L) | Before and after 1, 2, 4, 6, and 12 weeks of TH-substitution.
  The % of decrease of serum thyroid parameters TSH after 1, 2, 4, 6, and 12 weeks of TH-substitution.
Thyroglobulin (Tg; ng/mL) | Before and after 1, 2, 4, 6, and 12 weeks of TH-substitution
  The % of decrease of serum thyroid parameters Tg after 1, 2, 4, 6, and 12 weeks of TH-substitution.
  Tg is a precursor of T3 and T4 and is a measurement for remaining thyroid (cancer) cells. Tg-levels are affected by TSH and therefore, we expect by reducing TSH-levels to also reduce Tg levels. Consecutive Tg-measurements in this study act as a secondary measure for TH substitution. Since Tg-values between patients variable, we will use the % decrease instead of absolute values.
QoL in patients treated with L-T3 or L-T4 | Before and after 2, 6, and 12 weeks of TH-substitution
  Quality of life will be assessed using standardized QoL questionnaires for thyroid- and thyroid cancer patient reported outcome. Our aim is to compare improvement of hypothyroid symptoms after initiation of therapy, and evaluate whether sings of hyperthyroidism and possible overtreatment are present. We will use the European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 (core measure QoL questionnaire) in combination with the THYCA-QoL (additional thyroid cancer-specific part).
Heart rate (HR; bpm) | Before and after 6 and 12 weeks of TH-substitution
  Cardiovascular parameters will be assessed during visits to the outpatient clinic before initiation of TH-substitution (during hypothyroidism) and after 6 weeks of TH-treatment. Patients will be compared intra- and interindividually.
Blood pressure (BP; mmHg) | Before and after 6 and 12 weeks of TH-substitution
  Cardiovascular parameters will be assessed during visits to the outpatient clinic before initiation of TH-substitution (during hypothyroidism) and after 6 and 12 weeks of TH-treatment. Patients will be compared intra- and interindividually.

CONTACTS AND LOCATIONS:
Overall Officials: Wouter Zandee, MD/PhD, Principal Investigator — University Medical Center Groningen
Locations (2):
- Netherlands (2):
  - University Medical Center Groningen (UMCG), Groningen, Provincie Groningen
  - Radboud University Nijmegen, Nijmegen

IPD SHARING:
Plan to Share IPD: No
Handling of personal data complies with the General Data Protection Regulation (GDPR; in Dutch: De uitvoeringswet algemene verorderning gegevensbescherming [UAVG]). Encoded data will be kept for 15 years after closure of the study and can only be used for ancillary studies after strict approval of the study protocol by the project leader (dr. W. Zandee).